CLINICAL TRIAL: NCT00003305
Title: A Phase II Trial of Aminopterin in Adults and Children With Refractory Acute Leukemia Grant Application Title: A Phase II Trial of Aminopterin in Acute Leukemia
Brief Title: Aminopterin in Treating Patients With Refractory Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066248; ILEX-AMT-002/1997; UTSMC-AMT-002/1997; UTSMC-FDR001458; NCI-V99-1534
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Aminopterin; Leucovorin

INTERVENTIONS:
Drug: aminopterin
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminopterin in treating patients who have refractory leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of aminopterin in patients with refractory leukemia and minimal previous exposure to antifolate agents. II. Determine the antileukemic activity of aminopterin in adults and children with acute myelogenous and acute lymphoblastic leukemia for whom conventional therapy has failed. III. Confirm that aminopterin can be administered for four consecutive weeks when followed with minimal leucovorin calcium rescue and determine the minimal amount of leucovorin calcium required for each patient. IV. Confirm bioavailability data on oral aminopterin by performing limited sampling pharmacokinetics. V. Correlate blast uptake of aminopterin in vitro with clinical response.

OUTLINE: This is an open label study. Patients are stratified according to age and type of leukemia: Stratum I: Under 20 years old with acute lymphoblastic leukemia (ALL) in second or greater relapse Stratum II: Greater than 20 years old with ALL in first or greater relapse Stratum III: Patients of any age with acute myelogenous leukemia (AML) in first or greater relapse Patients receive aminopterin every 12 hours for 2 doses weekly for 4 weeks. Aminopterin is administered intravenously over 20 minutes for the first, second, and fourth doses, and orally for the third dose. The fifth and all subsequent doses are administered orally if bioavailability is acceptable. Patients receive oral leucovorin calcium every 12 hours for 2 doses beginning 24 hours after the last dose of aminopterin each week. If toxicity is limited for 2 consecutive weeks, the dose of leucovorin calcium is decreased to 1 dose administered 24 hours after the last dose of aminopterin each week. If this schedule is tolerated for 2 consecutive weeks, then leucovorin calcium is discontinued. Patients continue therapy for up to 15 months in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months.

PROJECTED ACCRUAL: This study will accrue a maximum of 25 patients per stratum, for a total of 75 patients, within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven acute leukemia of any histologic type that is refractory to known effective therapy

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 50-100% Life expectancy: At least 6 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL ALT no greater than 5 times upper limit of normal Renal: Creatinine normal for age Cardiovascular: No unstable angina No uncontrolled arrhythmia Pulmonary: No third space effusion Other: No severe uncontrolled infection Adequate nutritional status At least third percentile for weight Normal total serum protein Normal albumin/globulin ratio No serious concurrent physical or mental illness Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior bone marrow transplantation Recovered from prior biologic therapy No concurrent anticancer biologic therapy Chemotherapy: Recovered from prior chemotherapy No concurrent anticancer chemotherapy Endocrine therapy: Recovered from prior endocrine therapy No concurrent anticancer endocrine therapy No concurrent dexamethasone or other steroids as antiemetic agents Radiotherapy: No concurrent anticancer radiotherapy Surgery: Not specified Other: No concurrent dairy products for 2-4 hours before, during, or 2-4 hours after study drug No concurrent trimethoprim-sulfamethoxazole or dapsone as prophylaxis for Pneumocystis infection No concurrent multivitamins containing folic acid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1997-07; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton A. Kamen, MD, PhD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (14):
- United States (14):
  - Advanced Urology Medical Center, Anaheim, California
  - South Coast Urological Medical Group, Laguana Hills, California
  - Urology Specialists, P.C., Waterbury, Connecticut
  - Barzell, Whitmore, Treiman and Dunne - The Urology Treatment Center, Sarasota, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - 206 Research Associates, Greenbelt, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Medical & Clinical Research Associates, LLC, Bay Shore, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Medical City Dallas Hospital, Dallas, Texas
  - Urology Centers of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Cole PD, Drachtman RA, Masterson M, Smith AK, Glod J, Zebala JA, Lisi S, Drapala DA, Kamen BA. Phase 2B trial of aminopterin in multiagent therapy for children with newly diagnosed acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2008 Jun;62(1):65-75. doi: 10.1007/s00280-007-0576-7. Epub 2007 Sep 2. PMID 17768625